CLINICAL TRIAL: NCT06506916
Title: A Phase 3b Exploratory Multicenter Open-Label Study to Evaluate the Effect of Bimekizumab on Gene Expression Biomarkers in Study Participants With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Effect of Bimekizumab on Gene Expression Biomarkers in Study Participants With Moderate to Severe Plaque Psoriasis
Acronym: BE UNIQUE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PS0039; 2023-506333-29-00 (Registry Identifier: EU Clinical Trials); U1111-1299-2563 (Other: World Health Organization)
Record Dates: First submitted 2024-07-09; First posted 2024-07-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Moderate to Severe Plaque Psoriasis; Psoriatic Arthritis
Keywords: Moderate to Severe Plaque Psoriasis; PSO; Phase 3; Bimekizumab; Biomarkers; PsA
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Study participants with moderate to severe plaque PSO without concomitant active PsA (Cohort A) receive bimekizumab dosage regimen 1 from Baseline up to Week 16 and bimekizumab regimen 2 from Week 16 up to Week 48. Study participants, fulfilling randomization criteria receive bimekizumab dosage regimen 2 or 3 from Week 48 to Week 96. Study participants who do not meet the criteria for randomization receive bimekizumab dosage regimen 2 to Week 96.
  Interventions: Drug: bimekizumab
- Cohort B (Experimental): Study participants with moderate to severe plaque PSO with concomitant active PsA (Cohort B) receive bimekizumab dosage regimen 1 from Baseline up to Week 16 and bimekizumab regimen 2 from Week 16 up to Week 48. Study participants, fulfilling randomization criteria receive bimekizumab dosage regimen 2 or 3 from Week 48 to Week 96. Study participants who do not meet the criteria for randomization receive bimekizumab dosage regimen 2 to Week 96.
  Interventions: Drug: bimekizumab
- Control Cohort (No Intervention): Healthy participants, who will not receive IMP during the study.

INTERVENTIONS:
Drug: bimekizumab — Study participants receive bimekizumab (BKZ) administered subcutaneously at pre-specified timepoints during study.
  Other Names: BKZ
  Arms: Cohort A; Cohort B

SUMMARY:
The purpose of this study is to evaluate the effect of bimekizumab on gene expression biomarkers at Week 48 in a subset of study participants with moderate to severe plaque psoriasis (PSO) and moderate to severe plaque PSO with concomitant active psoriatic arthritis (PsA) who have provided skin biopsies for reverse transcription-polymerase chain reaction (RT-PCR).

ELIGIBILITY:
Inclusion Criteria:

Cohort A and Cohort B

* Study participant must be at least 18 years of age inclusive at the time of signing the Informed Consent Form (ICF)
* Study participant must have:

  1. Cohort A and Cohort B: Plaque psoriasis (PSO) diagnosed for at least 6 months prior to the Screening Visit
  2. Cohort B only: In addition to the criteria specified above, study participant has a documented diagnosis of adult-onset psoriatic arthritis (PsA) and meets the CASPAR classification criteria for at least 6 months prior to Screening for active PsA and must have ≥1 tender joint count (TJC) out of 68 and ≥1 swollen joint count (SJC) out of 66 at Screening or up to 3 months before Screening (documented evidence)
* Study participant must have Psoriasis Area and Severity Index (PASI) score ≥12 and body surface area (BSA) affected by PSO ≥10% and Investigator's Global Assessment (IGA) score ≥3 on a 5 point scale
* Study participant must be a candidate for systemic PSO therapy and/or phototherapy
* Study participant agrees not to change their usual sun exposure during the course of the study and to use ultraviolet A/ultraviolet B sunscreens if unavoidable exposure occurs
* Study participant has body weight <120 kg
* A female study participant is eligible to participate if they are not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the Run In Treatment Period, the Randomized Treatment Extension Period, theTreatment Extension Period, the Escape Treatment Period, and for 17 weeks after the final dose of investigational medicinal product (IMP)

Control Cohort

* Study participant must be ≥18 years of age at the time of signing the informed consent
* Study participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and vital signs
* Study participant has body weight <120 kg
* Female study participant is eligible to participate if they are not pregnant and not breastfeeding

Exclusion Criteria:

Cohort A and Cohort B

* Study participant has a form of PSO other than plaque type (eg, pustular, erythrodermic and guttate PSO, or drug induced PSO)
* Study participant has an active infection or history of infection(s) as follows:

  1. Any active systemic infection within 14 days prior to Baseline
  2. A serious infection, defined as requiring hospitalization or intravenous anti-infective(s) within 2 months prior to the Baseline Visit
  3. A history of opportunistic, recurrent, or chronic infections that, in the opinion of the investigator, might cause this study to be detrimental to the study participant
* At investigator's discretion, study participant with chronic (medically controlled) viral hepatitis B or C or human immunodeficiency virus (HIV) infection, or history of hepatitis B.
* Study participant has any of the following:

  1. Known active tuberculosis (TB) disease.
  2. History of active TB involving any organ system unless adequately treated
  3. High risk of acquiring TB infection
* Study participant has a verified diagnosis of inflammatory conditions other than PSO or PsA, including but not limited to rheumatoid arthritis (RA), sarcoidosis, inflammatory bowel diseases (IBD), or systemic lupus erythematosus. Note: Study participants with a diagnosis of IBD are allowed if they have no active symptomatic disease at Screening or Baseline
* Study participant has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer
* Study participant has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Study participant has a known hypersensitivity to any components of the IMP as stated in this protocol
* Study participant has a history of primary failure to any biologic (ie, no response within the first 12 weeks of treatment)
* Study participant has laboratory abnormalities at Screening
* Study participant has a current history of alcohol or drug use disorder, as defined in Diagnostic and Statistical Manual of Mental Disorders (DSM) V, within the previous 6 months prior to Screening, as evaluated by the investigator based on medical history, and/or site interview

Control Cohort

- Study participant has any systemic disease (eg, cardiovascular, neurological, renal, liver, metabolic, gastrointestinal, hematological, coagulation disorders, immunological) considered by the investigator to be uncontrolled, unstable, or likely to progress to a clinically significant degree during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2027-03-09 (Estimated); Study Completion 2028-03-14 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in composite gene expression score using reverse transcription-polymerase chain reaction (RT-PCR) in lesional skin at Week 48 | Week 48, compared to Baseline
  Composite gene expression score using RT-PCR in lesional skin at Baseline and Week 48 using preselected genes based on bimekizumab mechanism of action and PSO disease biology pathways.

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) from Baseline to the end of the Safety Follow-Up (SFU) | From Baseline to End of SFU (up to Week 100)
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. TEAEs are defined as those AEs that have a start date on or following the first dose of IMP through SFU (at least 12 weeks after final IMP dose and not before 4 weeks after the last skin biopsy).
Treatment-emergent serious adverse event (TESAEs) from Baseline to the end of the SFU | From Baseline to End of SFU (up to Week 100)
  A serious adverse event (SAE) must meet 1 or more of the following criteria:
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent disability/incapacity
  * Is a congenital anomaly/birth defect
  * Important medical event that, based upon appropriate medical judgment, may jeopardize the patient or subject and may require medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious.
  TESAEs are defined as those SAEs that have a start date on or following the first dose of IMP through SFU (at least 12 weeks after final IMP dose and not before 4 weeks after the last skin biopsy).
TEAEs leading to permanent discontinuation of IMP from Baseline to the end of the SFU | From Baseline to End of SFU (up to Week 100)
  This measure considers any TEAE leading to permanent discontinuation of IMP regardless of reason.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (16):
- United States (7):
  - Ps0039 50140, Birmingham, Alabama
  - Ps0039 50162, Fountain Valley, California
  - Ps0039 50642, Santa Monica, California
  - Ps0039 50283, Tampa, Florida
  - Ps0039 50110, Ann Arbor, Michigan
  - Ps0039 50643, Rochester, New York
  - Ps0039 50491, Pittsburgh, Pennsylvania
- Germany (4):
  - Ps0039 40515, Berlin
  - Ps0039 40287, Frankfurt am Main
  - Ps0039 40072, Freiburg im Breisgau
  - Ps0039 40775, Witten
- Poland (5):
  - Ps0039 40347, Lodz
  - Ps0039 40625, Lodz
  - Ps0039 40757, Poznan
  - Ps0039 40761, Warsaw
  - Ps0039 40773, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if a determination is made that the data cannot be adequately anonymized.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://Vivli.org